CLINICAL TRIAL: NCT05272787
Title: A Single-Center, Open-Label, Randomized Safety-in-Use Clinical Study to Assess the Topical Tolerability and Efficacy of a Facial Moisturizer and Lip Moisturizer During and After 21±2 Days of Use in Adult Subjects Undergoing a Facial Dermatologic Procedure With Fractional CO2 Laser
Brief Title: Clinical Trial to Evaluate Safety and Efficacy of a Facial and Lip Moisturizer in Adult Subjects Undergoing a Facial Dermatologic Procedure With Fractional CO2 Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCSSKA004711
Record Dates: First submitted 2022-02-25; First posted 2022-03-09 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Skin Regeneration After Dermatological Facial Procedure With Fractional CO2 Laser
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Intervention Model Description: All participants will receive the same study regimen consisting of 5 products: a facial moisturizer, a facial moisturizer (control), a lip moisturizer, a sunscreen and a facial wash.The facial moisturizers will be applied on the half face. The choice of the half face on which the product will be applied will be defined by a randomization list, prepared by the statistician in charge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left face TH Facial Moisturizer (Experimental): All subjects will receive all the products. There will be a supervised application at the site on the baseline visit of the study. Then subjects will use all the products at home. The choice of the half face on which the product will be applied will be defined by a randomization list, prepared by the statistician in charge. If the TH Facial Moisturizer will be applied on the left side of the face, then the Facial Moisturizer B (Control) will be applied on the right side of the face. Lip moisturizer, facial wash and sunscreen will be applied in all arms of the study.
  Interventions: Other: TH Facial Moisturizer; Other: TH Lip Moisturizer; Other: Facial Moisturizer B (Control); Other: Sunscreen; Other: Facial wash
- Right face TH Facial Moisturizer (Experimental): All subjects will receive all the products. There will be a supervised application at the site on the baseline visit of the study. Then subjects will use all the products at home. The choice of the half face on which the product will be applied will be defined by a randomization list, prepared by the statistician in charge. If the TH Facial Moisturizer will be applied on the right side of the face, then the Facial Moisturizer B (Control) will be applied on the left side of the face. Lip moisturizer, facial wash and sunscreen will be applied in all arms of the study.
  Interventions: Other: TH Facial Moisturizer; Other: TH Lip Moisturizer; Other: Facial Moisturizer B (Control); Other: Sunscreen; Other: Facial wash

INTERVENTIONS:
Other: TH Facial Moisturizer — All subjects will receive all the products. There will be a supervised application at the site on the baseline visit of the study. Then subjects will use all the products at home.
  Other Names: The Facial lotion product is a moisturizing formulation intended for topical use on the half-face. It will be applied at least twice daily.
Other: TH Lip Moisturizer — All subjects will receive all the products. There will be a supervised application at the site on the baseline visit of the study. Then subjects will use all the products at home.
  Other Names: The lip lotion product is a moisturizing formulation intended for topical use on the lips. It will be applied at least twice daily.
Other: Facial Moisturizer B (Control) — All subjects will receive all the products. There will be a supervised application at the site on the baseline visit of the study. Then subjects will use all the products at home.
  Other Names: The Facial lotion product is a moisturizing formulation intended for topical use on the half-face. It will be applied at least twice daily.
Other: Sunscreen — Auxiliary product
  Other Names: It will be used all over the face whenever there is the intention of sun exposure.
Other: Facial wash — Auxiliary product.
  Other Names: It will be used to wash the face at least once daily.

SUMMARY:
This is study aims to evaluate the topical safety (tolerability/acceptability) and efficacy of TH Facial Moisturizer and TH Lip Moisturizer Investigational products after 21 ± 2 days of use under normal conditions on the half-face by adult participants who underwent dermatological facial procedure with fractional CO2 Laser under the supervision of a dermatologist. For these investigational products, safety parameters, clinical efficacy, instrumental efficacy (skin hydration, skin barrier integrity and facial imaging) and perceived efficacy through subjective perception questionnaires will be evaluated. Subjects will receive the product to use it at home for 21 +/- 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or Female
* 18 to 65 years old
* Fitzpatrick Skin Type I to III
* Generally in good health based on medical history reported by the subject.
* Subjects presenting dry/dried up lips, proven by dermatologist.
* Subjects who have some cutaneous condition whose performance of the Fractional CO2 Laser procedure is recommended by the dermatologist, for example facial spots and/or acne scars and/or facial wrinkles.
* Able to read, write, speak, and understand Portuguese.
* Individual has signed the ICD.
* Agree to the performance of the Fractional CO2 Laser procedure by the dermatologist.
* Agree to use two facial products, each on one half face, and one lip product.
* Agree to use the facial sunscreen provided during the conditioning period and during sun exposure.
* Agree to replace their usual facial wash with the facial wash provided for facial cleansing during the conditioning period and during the study.
* For male participants: agree to shave the day before visits 2, 4 and 5.
* Intends to complete the study and is willing and able to follow all study instructions.

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products including facial moisturizer, sunscreen and liquid soap.
* Have known allergies or adverse reactions to the Pliaglis anesthetic cream that will be used for the dermatological facial procedure.
* Presents with a skin condition that may confound the study results (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer).
* Presents with primary/secondary lesions (scar - except from acne, ulcers, vesicles) or tattoos on test sites.
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication.
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:
* Immunosuppressive or steroidal drugs within 2 months before Visit 1*
* Non-steroidal anti-inflammatory drugs within 5 days before Visit 1*
* Antihistamines within 2 weeks before Visit 1*

  * If an individual is taking one of these medication types, the individual is not considered eligible at screening. However, if a subject begins using one of these medications during the study, the Study Physician should be consulted to consider the impact of the specific medication on subject safety and/or the study results, as described in section "Concurrent/Concomitant Medication".
* Is self-reported to be pregnant or planning to become pregnant during the study.
* Subjects with a history of keloid formation.
* Subject with a history of Herpes.
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study.
* Test positive for COVID-19 at visit 2 according to the rapid antigen test (COVID-19 Ag Immuno-Rapid Kit).
* Is simultaneously participating in any other clinical study.
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor.
* History of a confirmed COVID-19 infection in the last 30 days.
* Contact with COVID-19-infected person within 14 days prior to all on-site visits.
* Any international travel within 14 days prior to all on-site visits including members in the same household.
* Subjects with self-reported symptoms within the past 2 weeks:
* Unexplained cough, shortness of breath/difficulty breathing, fatigue, body aches (headaches, muscle pain, stomach aches), conjunctivitis, loss of smell, loss of taste, poor appetite, nausea, vomiting, diarrhea, palpitations, fever, or chest pain/tightness.
* Temperature ≥ 38.0°C /100.4°F, measured.
* Use of fever reducers within the past 2 days of each onsite visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline of scores of erythema to 21 ± 2 days. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole face (including lips) and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole face (including lips). The change from baseline will be evaluated to assess skin tolerance of the TH Facial moiturizer and TH Lip moisturizer.
Change from baseline of the scores of desquamation to 21 ± 2 days. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole face (including lips) and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole face (including lips). The change from baseline will be evaluated to assess skin tolerance of the TH Facial moiturizer and TH Lip moisturizer.
Change from baseline of the scores of blistering to 21 ± 2 days. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole face (including lips) and score the identified blisterings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole face (including lips). The change from baseline will be evaluated to assess skin tolerance of the TH Facial moiturizer and TH Lip moisturizer.
Change from baseline of the scores of edema to 21 ± 2 days. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the whole face (including lips) and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify this skin reaction on the whole face (including lips). The change from baseline will be evaluated to assess skin tolerance of the TH Facial moiturizer and TH Lip moisturizer.
Percentage of participants with Adverse Events through 21 ± 2 days. | 21 ± 2 days.
  The percentage of participants with AEs, serious adverse events (SAEs), AEs leading to discontinuation and AEs related to skin reactions will be evaluated for skin tolerance up to 21 ± 2 days.

SECONDARY OUTCOMES:
Change from baseline of the scores of erythema to 21 ± 2 days for TH facial moisturizer. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of erythema to 21 ± 2 days for Facial Moisturizer B (Control). | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of erythema scores at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | 21 ± 2 days.
  At 21 ± 2 days, the study physician will evaluate both half faces and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 21 ± 2 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of erythema to 5 ± 1 day for TH facial moisturizer. | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of erythema to 5 ± 1 day for Facial Moisturizer B (Control). | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of erythema scores at5 ± 1 day between TH facial moisturizer and Facial Moisturizer B (Control) | At 5 ± 1 day.
  At 5 ± 1 day, the study physician will evaluate both half faces and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 5 ± 1 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of erythema to 24 hours for TH facial moisturizer. | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of erythema to 24 hours for Facial Moisturizer B (Control). | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of erythema scores at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the study physician will evaluate both half faces and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 24 hours scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of erythema to 1 hour for TH facial moisturizer. | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of erythema to 1 hour for Facial Moisturizer B (Control). | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of erythema scores at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the study physician will evaluate both half faces and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 1-hour scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of erythema to 30 minutes for TH facial moisturizer. | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of erythema to 30 minutes for Facial Moisturizer B (Control). | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of erythema scores at 30 minutes between TH facial moisturizer and Facial Moisturizer B (Control) | At 30 minutes.
  At 30 minutes, the study physician will evaluate both half faces and score the identified erythemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 30 minutes scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of edema to 21 ± 2 days for TH facial moisturizer. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of edema to 21 ± 2 days for Facial Moisturizer B (Control). | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of edema scores at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, the study physician will evaluate both half faces and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 21 ± 2 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of edema to 5 ± 1 day for TH facial moisturizer. | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of edema to 5 ± 1 day for Facial Moisturizer B (Control). | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of edema scores at 5 ± 1 day between TH facial moisturizer and Facial Moisturizer B (Control) | At 5 ± 1 day.
  At 5 ± 1 day, the study physician will evaluate both half faces and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 5 ± 1 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of edema to 24 hours for TH facial moisturizer. | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of edema to 24 hours for Facial Moisturizer B (Control). | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of edema scores at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the study physician will evaluate both half faces and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 24 hours scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of edema to 1 hour for TH facial moisturizer. | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of edema to 1 hour for Facial Moisturizer B (Control). | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of edema scores at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the study physician will evaluate both half faces and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 1-hour scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of edema to 30 minutes for TH facial moisturizer. | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of edema to 30 minutes for Facial Moisturizer B (Control). | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of edema scores at 30 minutes between TH facial moisturizer and Facial Moisturizer B (Control) | At 30 minutes.
  At 30 minutes, the study physician will evaluate both half faces and score the identified edemas according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 30 minutes scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of dryness to 21 ± 2 days for TH facial moisturizer. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of dryness to 21 ± 2 days for Facial Moisturizer B (Control). | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of dryness scores at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, the study physician will evaluate both half faces and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 21 ± 2 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of dryness to 5 ± 1 day for TH facial moisturizer. | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of dryness to 5 ± 1 day for Facial Moisturizer B (Control). | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of dryness scores at 5 ± 1 day between TH facial moisturizer and Facial Moisturizer B (Control) | At 5 ± 1 day.
  At 5 ± 1 day, the study physician will evaluate both half faces and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 5 ± 1 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of dryness to 24 hours for TH facial moisturizer. | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of dryness to 24 hours for Facial Moisturizer B (Control). | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of dryness scores at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the study physician will evaluate both half faces and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 24 hours scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of dryness to 1 hour for TH facial moisturizer. | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of dryness to 1 hour for Facial Moisturizer B (Control). | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of dryness scores at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the study physician will evaluate both half faces and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 1-hour scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of dryness to 30 minutes for TH facial moisturizer. | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of dryness to 30 minutes for Facial Moisturizer B (Control). | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of dryness scores at 30 minutes between TH facial moisturizer and Facial Moisturizer B (Control) | At 30 minutes.
  At 30 minutes, the study physician will evaluate both half faces and score the identified dryness according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 30 minutes scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of desquamation to 21 ± 2 days for TH facial moisturizer. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of desquamation to 21 ± 2 days for Facial Moisturizer B (Control). | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of desquamation scores at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, the study physician will evaluate both half faces and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 21 ± 2 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of desquamation to 5 ± 1 day for TH facial moisturizer. | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of desquamation to 5 ± 1 day for Facial Moisturizer B (Control). | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of desquamation scores at 5 ± 1 day between TH facial moisturizer and Facial Moisturizer B (Control) | At 5 ± 1 day.
  At 5 ± 1 day, the study physician will evaluate both half faces and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 5 ± 1 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of desquamation to 24 hours for TH facial moisturizer. | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of desquamation to 24 hours for Facial Moisturizer B (Control). | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of desquamation scores at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the study physician will evaluate both half faces and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 24 hours scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of desquamation to 1 hour for TH facial moisturizer. | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of desquamation to 1 hour for Facial Moisturizer B (Control). | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of desquamation scores at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the study physician will evaluate both half faces and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 1-hour scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of desquamation to 30 minutes for TH facial moisturizer. | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of desquamation to 30 minutes for Facial Moisturizer B (Control). | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of desquamation scores at 30 minutes between TH facial moisturizer and Facial Moisturizer B (Control) | At 30 minutes.
  At 30 minutes, the study physician will evaluate both half faces and score the identified desquamations according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 30 minutes scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of stinging to 21 ± 2 days for TH facial moisturizer. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of stinging to 21 ± 2 days for Facial Moisturizer B (Control). | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of stinging scores at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, the study physician will evaluate both half faces and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 21 ± 2 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of stinging to 5 ± 1 day for TH facial moisturizer. | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of stinging to 5 ± 1 day for Facial Moisturizer B (Control). | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of stinging scores at 5 ± 1 day between TH facial moisturizer and Facial Moisturizer B (Control) | At 5 ± 1 day.
  At 5 ± 1 day, the study physician will evaluate both half faces and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 5 ± 1 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of stinging to 24 hours for TH facial moisturizer. | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of stinging to 24 hours for Facial Moisturizer B (Control). | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of stinging scores at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the study physician will evaluate both half faces and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 24 hours scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of stinging to 1 hour for TH facial moisturizer. | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of stinging to 1 hour for Facial Moisturizer B (Control). | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of stinging scores at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the study physician will evaluate both half faces and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 1-hour scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of stinging to 30 minutes for TH facial moisturizer. | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of stinging to 30 minutes for Facial Moisturizer B (Control). | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of stinging scores at 30 minutes between TH facial moisturizer and Facial Moisturizer B (Control) | At 30 minutes.
  At 30 minutes, the study physician will evaluate both half faces and score the identified stingings according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 30 minutes scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of itching to 21 ± 2 days for TH facial moisturizer. | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of itching to 21 ± 2 days for Facial Moisturizer B (Control). | 21 ± 2 days.
  At baseline and at 21 ± 2 days, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of itching scores at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, the study physician will evaluate both half faces and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 21 ± 2 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of itching to 5 ± 1 day for TH facial moisturizer. | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of itching to 5 ± 1 day for Facial Moisturizer B (Control). | 5 ± 1 day.
  At baseline and at 5 ± 1 day, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of itching scores at 5 ± 1 day between TH facial moisturizer and Facial Moisturizer B (Control) | At 5 ± 1 day.
  At 5 ± 1 day, the study physician will evaluate both half faces and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 5 ± 1 day scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of itching to 24 hours for TH facial moisturizer. | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of itching to 24 hours for Facial Moisturizer B (Control). | 24 hours.
  At baseline and at 24 hours, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of itching scores at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the study physician will evaluate both half faces and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 24 hours scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of itching to 1 hour for TH facial moisturizer. | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of itching to 1 hour for Facial Moisturizer B (Control). | 1 hour.
  At baseline and at 1 hour, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of itching scores at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the study physician will evaluate both half faces and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 1-hour scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Change from baseline of the scores of itching to 30 minutes for TH facial moisturizer. | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the TH Facial moisturizer.
Change from baseline of the scores of itching to 30 minutes for Facial Moisturizer B (Control). | 30 minutes.
  At baseline and at 30 minutes, the study physician will evaluate the corresponding half face and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on the corresponding half face. The change from baseline will be evaluated to assess the clinical efficacy of the Facial Moisturizer B (Control).
Comparison of itching scores at 30 minutes between TH facial moisturizer and Facial Moisturizer B (Control) | At 30 minutes.
  At 30 minutes, the study physician will evaluate both half faces and score the identified itching according to the following intensity scale: 0 (absent); 1 (mild); 2 (moderate); 3 (intense).
  This scale will be used to classify the clinical evaluation on each half face. The 30 minutes scores of each half face will be compared with each other to compare the clinical efficacy of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Self-Perceived Efficacy Questionnaire at 30 minutes | 30 minutes
  Perceived efficacy related to the product usage will be subjectively evaluated by the participants through a questionnaire with questions related to use of the TH facial moisturizer and TH lip moisturezer produts. Participants will answer each question using a qualitative scale (agreement scale).
  This questionnaire will be used to evaluate the efficacy of TH Facial Moisturizing and TH Lip Moisturizer regarding skin regeneration after dermatological facial procedure with CO2 fractional laser in adult participants. The responses for each question will be provided as percentages.
Self-Perceived Efficacy Questionnaire at 24 hours | 24 hours
  Perceived efficacy related to the product usage will be subjectively evaluated by the participants through a questionnaire with questions related to use of the TH facial moisturizer and TH lip moisturezer produts. Participants will answer each question using a qualitative scale (agreement scale).
  This questionnaire will be used to evaluate the efficacy of TH Facial Moisturizing and TH Lip Moisturizer regarding skin regeneration after dermatological facial procedure with CO2 fractional laser in adult participants. The responses for each question will be provided as percentages.
Self-Perceived Efficacy Questionnaire at 5 ± 1 day | 5 ± 1 day
  Perceived efficacy related to the product usage will be subjectively evaluated by the participants through a questionnaire with questions related to use of the TH facial moisturizer and TH lip moisturezer produts. Participants will answer each question using a qualitative scale (agreement scale).
  This questionnaire will be used to evaluate the efficacy of TH Facial Moisturizing and TH Lip Moisturizer regarding skin regeneration after dermatological facial procedure with CO2 fractional laser in adult participants. The responses for each question will be provided as percentages.
Self-Perceived Efficacy Questionnaire at 21 ± 2 days | 21 ± 2 days
  Perceived efficacy related to the product usage will be subjectively evaluated by the participants through a questionnaire with questions related to use of the TH facial moisturizer and TH lip moisturizer products. Participants will answer each question using a qualitative scale (agreement scale).
  This questionnaire will be used to evaluate the efficacy of TH Facial Moisturizing and TH Lip Moisturizer regarding skin regeneration after dermatological facial procedure with CO2 fractional laser in adult participants. The responses for each question will be provided as percentages.
Visual skin condition of the whole face at baseline captured photographically | baseline
  Face images will be captured using a recognized device (Visia CR) at baseline to visualize the skin condition of these areas after the dermatological facial procedure with CO2 fractional laser and before the TH Facial moisturizer and Facial Moisturizer B (Control) usage on each determined half face.
  No analysis is planned. These images will be used as a qualitative complement to the other results for TH Facial moisturizer.
Visual skin condition of the whole face at 1 hour captured photographically | 1 hour
  Face images will be captured using a recognized device (Visia CR) at 1 hour to visualize the skin condition of these areas after the TH Facial moisturizer and Facial Moisturizer B (Control) supervised application on each determined half face.
  No analysis is planned. These images will be used as a qualitative complement to the other results for TH Facial moisturizer.
Visual skin condition of the whole face at 24 hours captured photographically | 24 hours
  Face images will be captured using a recognized device (Visia CR) at 24 hours to visualize the skin condition of these areas after the TH Facial moisturizer and Facial Moisturizer B (Control) usage on each determined half face.
  No analysis is planned. These images will be used as a qualitative complement to the other results for TH Facial moisturizer.
Visual skin condition of the whole face at 5 ± 1 day captured photographically | 5 ± 1 day
  Face images will be captured using a recognized device (Visia CR) at 5 ± 1 day to visualize the skin condition of these areas after the TH Facial moisturizer and Facial Moisturizer B (Control) usage on each determined half face.
  No analysis is planned. These images will be used as a qualitative complement to the other results for TH Facial moisturizer.
Visual skin condition of the whole face at 21 ± 2 days captured photographically | 21 ± 2 days
  Face images will be captured using a recognized device (Visia CR) at 21 ± 2 days to visualize the skin condition of these areas after the TH Facial moisturizer and Facial Moisturizer B (Control) usage on each determined half face.
  No analysis is planned. These images will be used as a qualitative complement to the other results for TH Facial moisturizer.
Mean change from baseline to 21 ± 2 days in skin hydration level for TH facial moisturizer. | 21 ± 2 days
  Skin hydration level of the determined half face will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the TH facial moisturizer on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 21 ± 2 days of usage.
Mean change from baseline to 21 ± 2 days in skin hydration level for Facial Moisturizer B (Control). | 21 ± 2 days
  Skin hydration level of the determined half face will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the Facial Moisturizer B (Control) on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 21 ± 2 days of usage.
Comparison of skin hydration level at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, skin hydration level of both half faces will be measured with corneometer, a recognized device that determine the water content of stratum corneum.
  This measure will be used to determine the effect of both products on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 21 ± 2 days of usage. The 21 ± 2 days measures of each half face will be compared with each other to compare the skin hydration of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Mean change from baseline to 24 hours in skin hydration level for TH facial moisturizer. | 24 hours
  Skin hydration level of the determined half face will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the TH facial moisturizer on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 24 hours of usage.
Mean change from baseline to 24 hours in skin hydration level for Facial Moisturizer B (Control). | 24 hours
  Skin hydration level of the determined half face will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the Facial Moisturizer B (Control) on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 24 hours of usage.
Comparison of skin hydration level at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, skin hydration level of both half faces will be measured with corneometer, a recognized device that determine the water content of stratum corneum.
  This measure will be used to determine the effect of both products on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 24 hours of usage. The 24 hours measures of each half face will be compared with each other to compare the skin hydration of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Mean change from baseline to 1 hour in skin hydration level for TH facial moisturizer. | 1 hour
  Skin hydration level of the determined half face will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the TH facial moisturizer on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 1 hour of supervised application.
Mean change from baseline to 1 hour in skin hydration level for Facial Moisturizer B (Control). | 1 hour
  Skin hydration level of the determined half face will be measured with corneometer, a recognized device that determine the water content of stratum corneum. This measure will be used to determine the effect of the Facial Moisturizer B (Control) on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser 1 hour of supervised application.
Comparison of skin hydration level at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour
  At 1 hour, skin hydration level of both half faces will be measured with corneometer, a recognized device that determine the water content of stratum corneum.
  This measure will be used to determine the effect of both products on skin hydration of the study population who underwent the dermatological facial procedure with CO2 fractional laser 1 hour of supervised application. The 1-hour measures of each half face will be compared with each other to compare the skin hydration of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Mean change from baseline to 21 ± 2 days in transepidermal water loss (TEWL) to assess skin barrier integrity for TH facial moisturizer. | 21 ± 2 days
  Skin barrier integrity of the determined half face will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
  This measure will be used to determine the effect of the TH facial moisturizer on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 21 ± 2 days of usage.
Mean change from baseline to 21 ± 2 days in transepidermal water loss (TEWL) to assess skin barrier integrity for Facial Moisturizer B (Control). | 21 ± 2 days
  Skin barrier integrity of the determined half face will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
  This measure will be used to determine the effect of the Facial Moisturizer B (Control) on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 21 ± 2 days of usage.
Comparison of transepidermal water loss (TEWL) to assess skin barrier integrity at 21 ± 2 days between TH facial moisturizer and Facial Moisturizer B (Control) | At 21 ± 2 days.
  At 21 ± 2 days, the transepidermal water loss of both half faces will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
  This measure will be used to determine the effect of both products on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 21 ± 2 days of usage. The 21 ± 2 days measures of each half face will be compared with each other to compare the skin barrier integrity of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Mean change from baseline to 24 hours in transepidermal water loss (TEWL) to assess skin barrier integrity for TH facial moisturizer. | 24 hours
  This measure will be used to determine the effect of the TH facial moisturizer on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 24 hours of usage.
  Skin barrier integrity of the determined half face will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
Mean change from baseline to 24 hours in transepidermal water loss (TEWL) to assess skin barrier integrity for Facial Moisturizer B (Control). | 24 hours
  This measure will be used to determine the effect of the Facial Moisturizer B (Control) on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 24 hours of usage.
  Skin barrier integrity of the determined half face will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
Comparison of transepidermal water loss (TEWL) to assess skin barrier integrity at 24 hours between TH facial moisturizer and Facial Moisturizer B (Control) | At 24 hours.
  At 24 hours, the transepidermal water loss of both half faces will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
  This measure will be used to determine the effect of both products on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 24 hours of usage. The 24 hours measures of each half face will be compared with each other to compare the skin barrier integrity of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).
Mean change from baseline to 1 hour in transepidermal water loss (TEWL) to assess skin barrier integrity for TH facial moisturizer. | 1 hour
  This measure will be used to determine the effect of the TH facial moisturizer on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 1 hour of supervised application.
  Skin barrier integrity of the determined half face will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
Mean change from baseline to 1 hour in transepidermal water loss (TEWL) to assess skin barrier integrity for Facial Moisturizer B (Control). | 1 hour
  This measure will be used to determine the effect of the Facial Moisturizer B (Control) on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 1 hour of supervised application.
  Skin barrier integrity of the determined half face will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
Comparison of transepidermal water loss (TEWL) to assess skin barrier integrity at 1 hour between TH facial moisturizer and Facial Moisturizer B (Control) | At 1 hour.
  At 1 hour, the transepidermal water loss of both half faces will be measured with Tewameter, a recognized device that determine the transepidermal water loss. Lower levels of TEWL may be related to a more integrate skin barrier.
  This measure will be used to determine the effect of both products on skin barrier integrity of the study population who underwent the dermatological facial procedure with CO2 fractional laser after 1 hour of supervised application. The 1-hour measures of each half face will be compared with each other to compare the skin barrier integrity of one product with the other (TH facial moisturizer versus Facial Moisturizer B (Control)).

CONTACTS AND LOCATIONS:
Overall Officials: Mariane Martins Mosca, Bsc., Principal Investigator — Allergisa Pesquisa Dermato-Cosmetica LTDA
Locations (1):
- Allergisa Pesquisa Dermato-Cosmetica Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Petrov A. Efficiency of Carbon Dioxide Fractional Laser in Skin Resurfacing. Open Access Maced J Med Sci. 2016 Jun 15;4(2):271-6. doi: 10.3889/oamjms.2016.062. Epub 2016 May 24. PMID 27335599
- [Background] Krupa Shankar D, Chakravarthi M, Shilpakar R. Carbon dioxide laser guidelines. J Cutan Aesthet Surg. 2009 Jul;2(2):72-80. doi: 10.4103/0974-2077.58519. PMID 20808594
- [Background] Zahr AS, Kononov T, Sensing W, Biron JA, Gold MH. An open-label, single-site study to evaluate the tolerability, safety, and efficacy of using a novel facial moisturizer for preparation and accelerated healing pre and post a single full-face radiofrequency microneedling treatment. J Cosmet Dermatol. 2019 Feb;18(1):94-106. doi: 10.1111/jocd.12817. Epub 2018 Nov 19. PMID 30456804
- [Background] ASSOCIAÇÃO MÉDICA MUNDIAL. Declaração de Helsinque. Princípios Éticos para Pesquisa Médica Envolvendo Participantes Humanos.Princípios Éticos para Pesquisa Médica Envolvendo Participantes Humanos.
- [Background] BRASIL. Ministério da Saúde. RDC nº 466, de 12 de dezembro 2012. Aprova diretrizes e normas regulamentadoras de pesquisas envolvendo seres humanos.
- [Background] Canfield Scientific. Visia CR: Facial Imaging System for Clinical Research. The Measuring Principle.
- [Background] Courage + Khazaka electronic GmbH. Corneometer® CM 825. The Measuring Principle.
- [Background] Courage + Khazaka electronic GmbH. Tewameter® TM 300. The Measuring Principle.
- [Background] Courage + Khazaka electronic GmbH. Tewameter® TM Nano. The Measuring Principle.
- [Background] International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use.. ICH harmonized tripartite guideline: Guideline for Good Clinical Practice. J Postgrad Med. 2001 Jan-Mar;47(1):45-50. No abstract available. PMID 11590294
- [Background] OPAS. Organização Pan-Americana de Saúde. Boas Práticas Clínicas: Documento das Américas. IV Conferência Pan-Americana para Harmonização da Regulamentação Farmacêutica, 2005.
- [Background] WAMA Diagnóstica. Guia para o teste rápido de antígeno: Kit Imuno-Rápido COVID-19 Ag. 2021.